CLINICAL TRIAL: NCT00004085
Title: Phase I/II Trial of High-Dose Radioimmunotherapy With a 90Y-Humanized MN-14 Anti-Carcinoembryonic Antigen (CEA) Antibody for the Treatment of Stage IV Breast Cancer
Brief Title: Radioimmunotherapy Plus Peripheral Stem Cell Transplantation in Treating Patients With Stage IV Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Garden State Cancer Center at the Center for Molecular Medicine and Immunology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Robert M Sharkey, GSCC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067297; R35CA039841 (NIH); CMMI-C-041A-98; NCI-H99-0039; NCI-V99-1568
Record Dates: First submitted 1999-12-10; First posted 2004-04-15 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Filgrastim; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim — as prescribed by physician
Procedure: autologous bone marrow transplantation — 1-2 weeks prior to treatment
Procedure: peripheral blood stem cell transplantation — 1-2 weeks prior to treatment
Radiation: yttrium Y 90 monoclonal antibody MN-14 — intravenous infusion over 30 min, single dose

SUMMARY:
RATIONALE: Radiolabeled monoclonal antibodies can locate tumor cells and deliver tumor-killing substances to them. Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by radioimmunotherapy used to kill tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of radiolabeled monoclonal antibody therapy plus peripheral stem cell transplantation in treating patients who have stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose and dose-limiting toxicity of yttrium Y 90 monoclonal antibody MN-14 (Y90 MOAB MN-14) plus peripheral blood stem cell rescue in patients with stage IV breast cancer. II. Determine the pharmacokinetic profile of Y90 MOAB MN-14 in the blood, normal organs, and tumors of this patient population. III. Determine the antibody response to Y90 MOAB MN-14 in these patients. IV. Determine the antitumor effect of this regimen in these patients. V. Determine the radiation absorbed dose to normal organs and tumors.

OUTLINE: This is a dose-escalation, multicenter study. Patients receive filgrastim (G-CSF) subcutaneously (SC) with or without chemotherapy on days -28 to -14 and peripheral blood stem cell (PBSC) collection on days -14 to -11. If an adequate number of CD34+ cells are not harvested, bone marrow may be collected. Patients receive pretherapy imaging with indium In 111 monoclonal antibody MN-14 IV for up to 40 minutes on day -7 followed by whole body imaging on days -7 to 0. Patients receive yttrium Y 90 monoclonal antibody MN-14 (Y90 MOAB MN-14) IV for up to 40 minutes on day 0. PBSC or bone marrow is reinfused on days 6 to 14, depending on antibody clearance. Patients receive G-CSF SC or IV until blood counts recover. Cohorts of 3-6 patients receive escalating doses of Y90 MOAB MN-14 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Patients are followed weekly for 2 months, monthly for 6 months, and then every 6 months for 5 years.

PROJECTED ACCRUAL: A total of 24-30 patients will be accrued for this study within 2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven stage IV breast cancer Measurable disease after firstline or greater chemotherapy Evidence of CEA expression by: Serum CEA at least 10 ng/mL OR Positive immunostaining of primary or metastatic tumors with a CEA-specific antibody Positive imaging of at least 1 confirmed tumor by pre-therapy indium In 111 monoclonal antibody MN-14 No brain metastases Bone marrow biopsy prior to stem cell mobilization required to assess cellularity and tumor involvement Cellularity greater than 60% of normal Tumor involvement less than 25% Chromosome analysis of bone marrow aspirate (optional) No brain metastases Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 and over Sex: Not specified Menopausal status: Not specified Performance status: Karnofsky 70-100% OR ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: WBC at least 3,000/mm3 Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 2 mg/dL AST less than 2 times upper limit of normal (ULN) Renal: Creatinine less than 1.5 times ULN Cardiovascular: Cardiac ejection fraction greater than 50% by MUGA Pulmonary: DLCO greater than 70% of predicted FVC and FEV1 greater than 70% of predicted Other: Not pregnant Negative pregnancy test Fertile patients must use effective contraception No severe anorexia, nausea or vomiting, or urinary incontinence No other significant concurrent medical problem including severe psychiatric, epileptic, or diabetic disease No prisoners If received prior chimeric or humanized antibody (e.g., trastuzumab (Herceptin)), must not have allergy to yttrium Y 90 monoclonal antibody MN-14

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior peripheral blood stem cell rescue Chemotherapy: See Disease Characteristics At least 1 course of prior chemotherapy At least 4 weeks since prior chemotherapy No prior high-dose chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy No prior radiotherapy to more than 30% of red bone marrow Surgery: At least 4 weeks since prior major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 1998-05; Primary Completion 2002-05 (Actual)

PRIMARY OUTCOMES:
Safety | 12 weeks
  maximum tolerated dose

CONTACTS AND LOCATIONS:
Overall Officials: Jack D. Burton, MD, Study Chair — Garden State Cancer Center at the Center for Molecular Medicine and Immunology
Locations (3):
- United States (3):
  - Garden State Cancer Center, Belleville, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania